CLINICAL TRIAL: NCT07208890
Title: Methotrexate Iontophoresis Versus Methotrexate 1% Gel on Depigmentation in Vitiligo Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Ola Mohamed Elsayed Elgohary, Lecturer, Department of Physical Therapy for cardiopulmonary , Pharos University, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pharos university
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Vitiligo - Evaluation of Methotrexate Iontophoresis and Topical Methotrexate Gel as Localized Treatment Approache

STUDY DESIGN:
Intervention Model Description: This study follows a randomized, parallel-group design involving 30 patients with stable vitiligo. Participants are randomly assigned into two equal groups: one group receives methotrexate iontophoresis (experimental group), and the other applies topical methotrexate 1% gel (control group). Both groups are treated for 8 weeks, and outcomes are compared based on pigmentation improvement (VASI) and quality of life (VIS-22)
Who Masked: Participant
Masking Description: This study is an open-label trial; neither participants nor investigators are blinded to the assigned intervention due to the different nature of application methods (iontophoresis vs. topical gel). However, outcome assessment using VASI and VIS-22 scores will be performed by an independent dermatologist who is blinded to the treatment allocation to minimize assessment bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate Iontophoresis (Experimental): Methotrexate Iontophoresis (Experimental Group)
  Type: Experimental
  Description: Participants will receive methotrexate iontophoresis using a low-intensity electric current (5-10 mA) for 15 minutes per session over 8 weeks - once weekly for the first 4 weeks and then every two weeks for the next 4 weeks (total 6 sessions).
  Device/Intervention: Iontophoresis with methotrexate solution
  Goal: To enhance transdermal drug delivery and promote repigmentation with minimal systemic absorption
  Interventions: Device: Methotrexate Iontophoresis/a low-intensity electric current
- Topical Methotrexate 1% Ge (Active Comparator): Type: Active Comparator
  Description: Participants will apply methotrexate 1% gel topically to the affected skin areas twice daily for 8 consecutive weeks.
  Intervention: Topical methotrexate 1% gel
  Goal: To assess the efficacy and safety of topical methotrexate alone compared to iontophoretic delivery
  Interventions: Device: Methotrexate Iontophoresis/a low-intensity electric current

INTERVENTIONS:
Device: Methotrexate Iontophoresis/a low-intensity electric current — : Application of methotrexate solution via iontophoresis using a low-intensity electric current (5-10 mA) for 15 minutes per session, once weekly for 4 weeks, then biweekly for another 4 weeks
  Other Names: : Application of methotrexate solution via iontophoresis using a low-intensity electric current (5-10 mA) for 15 minutes per session, once weekly for 4 weeks, then biweekly for another 4 weeks

SUMMARY:
Vitiligo is a common autoimmune depigmenting disorder characterized by selective destruction of melanocytes. Methotrexate (MTX) has shown potential in stabilizing disease activity and promoting repigmentation; however, systemic administration may cause hepatotoxicity. This pilot study aims to compare the efficacy and safety of methotrexate iontophoresis versus topical methotrexate 1% gel in patients with vitiligo. Thirty patients will be randomly assigned into two equal groups: Group A will receive methotrexate iontophoresis (5-10 mA, 15 min/session) for 8 weeks, while Group B will apply methotrexate 1% gel twice daily for 8 weeks. Outcomes will be assessed using the Vitiligo Area and Severity Index (VASI) and the Vitiligo Impact Scale-22 (VIS-22), with liver function monitored monthly

DETAILED DESCRIPTION:
Vitiligo is an autoimmune depigmenting disorder characterized by melanocyte destruction. Methotrexate (MTX) has shown potential in modulating autoimmune activity and promoting repigmentation, but systemic use carries hepatotoxic risks. This pilot randomized study compares methotrexate iontophoresis and topical methotrexate 1% gel in stable vitiligo patients. Thirty participants will be assigned equally into two groups: the iontophoresis group will receive MTX via low-intensity electric current sessions for 8 weeks, while the control group will apply topical MTX gel twice daily for the same period. Efficacy will be evaluated using the Vitiligo Area and Severity Index (VASI) and quality of life by the Vitiligo Impact Scale-22 (VIS-22). Liver function will be monitored monthly to ensure safety

ELIGIBILITY:
Inclusion Criteria:Clinically diagnosed vitiligo confirmed by a dermatologist.

Stable vitiligo for at least 6 months (no new lesions or progression).

Age between 18 and 60 years.

Both male and female patients.

Presence of localized or segmental vitiligo suitable for topical treatment.

Willingness to avoid other vitiligo treatments (e.g., phototherapy, corticosteroids) during the study period.

Able and willing to provide written informed consent and comply with study procedures -

Exclusion Criteria:History of systemic or topical methotrexate use within the past 3 months.

Unstable or rapidly progressive vitiligo during the last 6 months.

Presence of other autoimmune or dermatologic disorders that could interfere with study evaluation (e.g., psoriasis, eczema, lupus).

Known hypersensitivity or allergy to methotrexate or any gel/iontophoresis components.

Hepatic, renal, or hematologic impairment (abnormal liver function or renal profile).

Pregnant or breastfeeding women, or those planning pregnancy during the study period.

Use of phototherapy, corticosteroids, or immunosuppressive therapy within the last 3 months.

Metal implants or pacemakers, which may contraindicate iontophoresis

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Vitiligo Area and Severity Index (VASI | 2 month
  in Vitiligo Area and Severity Index (VASI) from baseline to week 8 to evaluate the degree of repigmentation
Vitiligo Impact Scale-22 (VIS-22) | 2month
  quality of life measured by the Vitiligo Impact Scale-22 (VIS-22), percentage of repigmentation in target lesions, and the proportion of participants achieving ≥50% repigmentatio

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a small-scale pilot study, and data sharing is not planned at this stage. Summary results may be available upon request from the principal investigator